CLINICAL TRIAL: NCT05834465
Title: Efficacy Evaluation of Anterior Chamber Drainage in Patients for High Intraocular Pressure After Cataract Surgery
Brief Title: High Intraocular Pressure After Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Principal Investigator, Wenzhou Medical University
Other Study IDs: 20230301CTR
Record Dates: First submitted 2023-03-24; First posted 2023-04-28 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Cataract; Intraocular Pressure
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: After using a non-contact tonometer to measure, the intraocular pressure is reduced by 0-10mmHg.
- Group 2: After using a non-contact tonometer to measure, the intraocular pressure is reduced by 10-20mmHg.
- Group 3: After using a non-contact tonometer to measure, the intraocular pressure is reduced over 20mmHg.

SUMMARY:
Effectiveness of anterior chamber drainage on the structure of the anterior chamber, the position of the intraocular lens and the shape of the corneal incision in the early stage of cataract surgery with high intraocular pressure

DETAILED DESCRIPTION:
To explore the effect of different degrees of anterior chamber drainage on the structure of the anterior chamber, the position of the intraocular lens and the shape of the corneal incision in the early stage of cataract surgery with high intraocular pressure

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 60 years old who underwent simple age-related cataract surgery in Eye Hospital of Wenzhou Medical University, the operation was successful, and there were no intraoperative complications such as posterior capsule rupture;
2. Measurements were taken before and after drainage, and all data were complete ;
3. The patient agrees and accepts the study.

Exclusion Criteria:

1. Preoperative glaucoma, ocular hypertension, iritis, uveitis and other eye diseases, as well as other eye diseases and serious systemic diseases that may affect the prognosis of surgery, such as corneal lesions, vitreous volume blood, retinal detachment, poor blood sugar control in diabetes, etc.
2. Previous history of eye trauma, etc.
3. Cannot cooperate with the completion of intraocular pressure measurement and CASIA2 examination.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Included in Eye Hospital of Wenzhou Medical University for "phacoemulsification combined with intraocular lens implantation" 2 hours after using a non-contact tonometer (FT-1000, TOMEY, JAPAN) to check that the intraocular pressure exceeds 28mmHg accompanied by corneal edema, anterior chamber radiation and age-related cataract patients over 60 years of age is required.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The position of IOL through tilt (tilt in degree) | Two hours after cataract surgery (i.e. before anterior chamber drainage)
  Evaluation of the position of IOL through tilt (tilt in degree)
The position of IOL through decentration (decentration in millimeter) | Two hours after cataract surgery (i.e. before anterior chamber drainage)
  Evaluation of the position of IOL through decentration (decentration in millimeter)
The position of IOL through tilt (tilt in degree) | Immediately after anterior chamber drainage
  Evaluation of the position of IOL through tilt (tilt in degree)
The position of IOL through decentration (decentration in millimeter) | Immediately after anterior chamber drainage
  Evaluation of the position of IOL through decentration (decentration in millimeter)

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No